CLINICAL TRIAL: NCT04285333
Title: Analgesic Techniques Before Spinal Anesthesia for Hip Fracture Repair: Ultrasound Percapsular Nerve Group Block VS Fascia Iliaca Block
Brief Title: Ultrasound Percapsular Nerve Group Block VS Fascia Iliaca Block for Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Collaborators: Institut Kassab d'Orthopédie (Other)
Responsible Party: Principal Investigator, Olfa kaabachi, MD, Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE-IMKO 102/2019
Record Dates: First submitted 2020-02-09; First posted 2020-02-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hip Fracture; Analgesia; Acute Pain
Keywords: hip fracture; nerve block; spinal anesthesia; analgesia
MeSH Terms: conditions — Hip Fractures; Agnosia; Acute Pain

STUDY DESIGN:
Intervention Model Description: Prospective randomised single blinded study
Who Masked: Participant, Care Provider
Masking Description: all blocks were performed in a special area outside operating room by docters only implicated in performance assessement of block and not in patient care. Patients where after moved to operating room, care provider wil assess pain before spinal anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fascial iliaca (Active Comparator): : A linear high frequency ultrasound probe (10-15MHz) was placed in a transverse direction over the anterior thigh below the inguinal ligament. We identified the femoral artery and the iliacus muscle lateral to it, covered by the fascia iliaca. The needle was inserted in plane and a 22 gauge, 50 mm needle was advanced until the tips placed underneath the fascia iliaca. Following negative aspiration, the local anesthetic solution was injected in 5mL increments while observing for adequate fluid spread in this plane for a total volume of 20 mL of 1.5% Lidocaine
  Interventions: Procedure: fascia iliaca block
- Percapsular nerve group block (Experimental): A curvilinear low-frequency ultrasound probe (2-5MHz) was initially placed in a transverse plane over the anterior inferior iliac spine (AIIS) and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the iliopubic eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed. A 22-gauge, 100-mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic solution was injected in 5 mL increments while observing for adequate fluid spread in this plane for a total volume of 20 mL of 1.5% Lidocaine.
  Interventions: Procedure: percapsular nerve group block

INTERVENTIONS:
Procedure: fascia iliaca block — ultrasound guided block with 20 mL lidocaine 1.5%
  Other Names: BIF for hip fracture
  Arms: fascial iliaca
Procedure: percapsular nerve group block — ultrasound guided block with 20 mL lidocaine 1.5%
  Other Names: PENG block for hip fracture
  Arms: Percapsular nerve group block

SUMMARY:
Spinal anesthesia (SA) is a widely accepted anesthetic technique for hip fracture repair among elderly. Positioning for SA can be extremely painful. Effective management of pain is important for these patients comfort.

Fascia Iliaca block (FIB) and Femoral nerve blocks are commonly used for analgesia in hip fracture patients. However, they often provide a modest reduction in pain.

The Percapsular Nerve Group block (PENG Block) has the advantage that it covers the accessory obturator nerve.

Aim of the study: compare FIB with PENG prior to positioning hip fracture patients for standardized SA.

In a prospective randomized double blind we included 80 patients aged more than 65 years old, for whom pain was felt when raising the affected limb to 15 degrees. Patients were assigned to receive either ultrasound guided Fascia Iliaca block or Percapsular Nerve Group block using 20 mL Lidocaine 1.5% in both groups. We compared pain on positioning for spinal anesthesia using Verbal Rating Scale (VRS 0 = no pain , VRS 1 = mild pain, t 2= severe pain) for both groups. We also recorded different times to perfom block.

DETAILED DESCRIPTION:
The purpose of the study was to compare analgesis effect of Percapsula nerve group block to fascia iliaca block prior to positioning hip fracture patients for standardized SA. We included 80 patients reporting pain with Verbal Rating Scale at 2 when raising the affected limb to 15 degrees. All patients admitted to induction room, were given standard monitoring and we randomized to receive either: ultrasound fascia iliaca block using linear high frequency ultrasound probe (10-15MHz) placed in a transverse direction over the anterior thigh below the inguinal ligament. A 50 mm needle was advanced until the tips placed underneath the fascia iliaca and 20 mL 1.5% Lidocaine was injected or ultrasound Percapsula nerve group block A curvilinear using low-frequency ultrasound probe (2-5MHz) that was initially placed in a transverse plane over the anterior inferior iliac spine and then aligned with the pubic ramus by rotating the probe counter clockwise approximately 45 degrees. In this view, the iliopubic eminence , the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed and than a 100 mm needle was advanced to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly and 20 mL 1.5% Lidocaine.We compared pain on positioning for spinal anesthesia and also different time to realise both blocks.

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged ≥ 65 years old and undergoing hip fracture surgical repair under continuous spinal anesthesia (CSA).
* Patients for whom pain was felt when raising the affected limb to 15 degrees (VERBAL PAIN SCALE =2)

Exclusion Criteria:

* - ASA physical status ≥ 4.
* Impaired cognition or Dementia.
* Multiple fractures.
* Contraindication to regional anesthesia.
* Patient's disapproval.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
positioning pain | up to 30 minutes
  Verbal Rating Scale (VRS) [0=no pain ; 4=worst pain]

SECONDARY OUTCOMES:
Positioning Rating | up to 40 minutes
  verbal rating scale (VRS) [0=no pain ; 4=worst pain]
Imaging time | up to 10 minutes
  For the PENG block:the femoral artery, the anterior inferior iliac spine, the iliopubic eminence and the psoas tendon.
  For the FIB: the femoral artery, the iliacus muscle, the fascia iliaca and the fascia lata.
Puncture time | up to 10 minutes
  the time that stretches from the introduction of the needle until the end of the injection of local anesthetic
Performance time | up to 10 minutes
  the imaging time + time to puncture.
Number of punctures | up to 10 minutes
  the number of redirection of the needle after removing 2 cm.
pain 5 after block | up to 5 minutes
  verbal rating scale (VRS) [0=no pain ; 4=worst pain]
pain 10 after block | up to 10 minutes
  verbal rating scale (VRS) [0=no pain ; 4=worst pain]
pain 15 after block | up to 15 minutes
  verbal rating scale (VRS) [0=no pain ; 4=worst pain]
pain 20 after block | up to 20 minutes
  verbal rating scale (VRS) [0=no pain ; 4=worst pain]

CONTACTS AND LOCATIONS:
Overall Officials: khaireddine Raddaoui, MD, Principal Investigator — Tunis El Manar University
Locations (1):
- Institut Kassab D'Orthopedie, Tunis, Tunisia